CLINICAL TRIAL: NCT01218178
Title: BIcarbonato di Sodio e N-Acetilcisteina Nella Prevenzione Della Nefropatia da Mezzo di Contrasto Nell'infaRto mIocardico acutO(Registro BINARIO)
Brief Title: Sodium Bicarbonate and N-Acetylcysteine for Nephroprotection in Acute Myocardial Infarction
Acronym: BINARIO
Status: Completed | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: Policlinico Casilino ASL RMB (Other)
Responsible Party: Principal Investigator, Antonio Maria Leone, MD, PhD, Catholic University of the Sacred Heart
Other Study IDs: P/479/CE/2010
Record Dates: First submitted 2010-10-04; First posted 2010-10-11 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-03

CONDITIONS: Acute Myocardial Infarction; Acute Kidney Injury
Keywords: acute myocardial infarction; acute kidney injury; contrast induced nephropathy; primary PCI; sodium-bicarbonate; N-acetylcysteine
MeSH Terms: conditions — Acute Kidney Injury | interventions — Sodium Bicarbonate

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sodium bicarbonate plus NAC: Sodium bicarbonate plus NAC
  Interventions: Drug: Sodium bicarbonate plus NAC
- Saline hydration plus NAC: Saline hydration plus NAC
  Interventions: Drug: Saline hydration plus NAC

INTERVENTIONS:
Drug: Sodium bicarbonate plus NAC — 154 mEq/L sodium bicarbonate (infusion rate of 3 ml/Kg for 1 hour followed by 1 ml/Kg for 6 hours) plus NAC (1200 mg bid for 48 hours)
  Groups: Sodium bicarbonate plus NAC
Drug: Saline hydration plus NAC — 0.9% saline (1 ml/Kg for 12 hours) plus NAC (1200 mg bid for 48 hours)
  Groups: Saline hydration plus NAC

SUMMARY:
Contrast-induced nephropathy (CIN) represents a potential complication of diagnostic and therapeutic procedures in interventional cardiology, especially in the acute setting of primary PCI. The investigators will test the efficacy of sodium bicarbonate (NaHCO3) and N-acetylcysteine (NAC) on the prevention of acute events and CIN in patients with acute myocardial infarction.

DETAILED DESCRIPTION:
Introduction Contrast-induced nephropathy (CIN) represents a potential complication of diagnostic and therapeutic procedures in interventional cardiology. In the setting of elective procedures, the strategy of sodium bicarbonate (NaHCO3) and N-acetylcysteine (NAC) infusion has been shown to reduce the incidence of CIN in high-risk patients. The efficacy of this strategy has not been demonstrated in the case of primary percutaneous coronary intervention (PCI).

Aim of the study The aim is to assess the efficacy of the strategy of sodium bicarbonate 154mEq/l + glucose solution 5% (infusion rate: 3 mL • kg-1 • h-1 for 1 hour followed by 1 mL • kg-1 • h-1 for 6 hours) and NAC (1200 mg i.v. followed by 1200 mg bid for the next 48 hours) in reducing the incidence of CIN in patients with STEMI undergoing primary or rescue PCI. As control group, a population of STEMI patients treated with NAC (1200 mg i.v. followed by 1200 mg bid for the next 48 hours) + conventional hydration with saline solution 0.9% will be retrospectively enrolled. According to the common definition, CIN will be defined as increase of the level of serum creatinine >0,5 mg/dL and/or increase ≥25% serum creatinine and/or decrease ≥25% of the glomerular filtration rate (GFR) as calculated with the MDRD Modification of Diet in Renal Disease)formula at 48 hours after PCI compared with baseline value after primary PCI.

Study Design This is a two-center (Policlinico Gemelli and Policlinico Casilino, Rome, Italy), prospective, spontaneous (not sponsored) observational study.

Patient population

Inclusion criteria:

* Consecutive patients with ST-Segment Elevation Myocardial Infarction (STEMI) as diagnosed according to the ACC (American College of Cardiology) criteria:

  * ischemic symptoms;
  * ECG variations: ST-elevation (>0,05 mV) in two or more contiguous leads;
  * Increase of the biochemical markers of myocardial necrosis (troponin T, cTNT).
* Indication to urgent coronary angiography and primary or rescue PCI

Exclusion criteria:

* Patients with history of allergic reaction to NAC (Fluimucil, Zambon Group Spa, Milan, Italy)
* Chronic hemodialysis
* Age > 90 years

Study protocol Patients will be treated with 154 mEq/L of sodium bicarbonate and glucose 5% solution (infusion rate of 3 mL • kg-1 • h-1 for 1 hour followed by 1 mL • kg-1 • h-1 for 6 hours) plus NAC (1200 mg i.v. followed by 1200 mg bid for the next 48 hours). As control group, a population of STEMI patients treated with conventional hydration with saline solution 0,9% and NAC (1200 mg i.v. followed by 1200 mg bid for the next 48 hours) according to the common clinical practice of the Department of Cardiovascular Medicine of the Policlinico Agostino Gemelli and of Cardiology Department of the Policlinico Casilino will be retrospectively enrolled.

Endpoints:

Primary endpoint:

- Composite endpoint (death/need for dialysis/CIN)

Secondary endpoints:

* assessment of individual major adverse events (death, re-infarction, need for dialysis) during at 1, 6 and 12 months
* assessment of the incidence of CIN defined as increase of the level of serum creatinine >0,5 mg/dL and/or increase ≥25% serum creatinine and/or decrease ≥25% of the glomerular filtration rate (GFR) as calculated with the MDRD formula at 48 hours after PCI compared with baseline value.

ELIGIBILITY:
Inclusion Criteria:

* ST-Segment Elevation Myocardial Infarction (STEMI) as diagnosed according to the ACC (American College of Cardiology) criteria:
* ischemic symptoms;
* ECG variations: ST-elevation (>0,05 mV) in two or more contiguous leads;
* Increase of the biochemical markers of myocardial necrosis (troponin T, cTNT). • Indication to urgent coronary angiography and primary or rescue PCI

Exclusion Criteria:

* Patients with history of allergic reaction to NAC
* Chronic hemodialysis
* Age >= 90 years

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: • Consecutive patients admitted from ER of the Policlinico Agostino Gemelli and Casilino of Rome with a ST-Segment Elevation Myocardial Infarction undergoing urgent PCI
Sampling Method: Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2008-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
All cause mortality, contrast-induced nephropathy and need of dialysis. | 2010
  To test the efficacy of sodium bicarbonate plus N-acetylcysteine vs saline hydration plus N-acetylcysteine to reduce mortality and to prevent contrast-induced nephropathy in the setting of primary PCI.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Maria Leone, MD, PhD, Principal Investigator — Catholic University of the Sacred Heart, Rome
Locations (1):
- Policlinico Agostino Gemelli and Policlinico Casilino, Rome, Italy

REFERENCES:
- [Background] Levey AS, Bosch JP, Lewis JB, Greene T, Rogers N, Roth D. A more accurate method to estimate glomerular filtration rate from serum creatinine: a new prediction equation. Modification of Diet in Renal Disease Study Group. Ann Intern Med. 1999 Mar 16;130(6):461-70. doi: 10.7326/0003-4819-130-6-199903160-00002. PMID 10075613
- [Background] Merten GJ, Burgess WP, Gray LV, Holleman JH, Roush TS, Kowalchuk GJ, Bersin RM, Van Moore A, Simonton CA 3rd, Rittase RA, Norton HJ, Kennedy TP. Prevention of contrast-induced nephropathy with sodium bicarbonate: a randomized controlled trial. JAMA. 2004 May 19;291(19):2328-34. doi: 10.1001/jama.291.19.2328. PMID 15150204
- [Background] Mehran R, Aymong ED, Nikolsky E, Lasic Z, Iakovou I, Fahy M, Mintz GS, Lansky AJ, Moses JW, Stone GW, Leon MB, Dangas G. A simple risk score for prediction of contrast-induced nephropathy after percutaneous coronary intervention: development and initial validation. J Am Coll Cardiol. 2004 Oct 6;44(7):1393-9. doi: 10.1016/j.jacc.2004.06.068. PMID 15464318
- [Background] Wright RS, Reeder GS, Herzog CA, Albright RC, Williams BA, Dvorak DL, Miller WL, Murphy JG, Kopecky SL, Jaffe AS. Acute myocardial infarction and renal dysfunction: a high-risk combination. Ann Intern Med. 2002 Oct 1;137(7):563-70. doi: 10.7326/0003-4819-137-7-200210010-00007. PMID 12353943
- [Background] Marenzi G, Lauri G, Assanelli E, Campodonico J, De Metrio M, Marana I, Grazi M, Veglia F, Bartorelli AL. Contrast-induced nephropathy in patients undergoing primary angioplasty for acute myocardial infarction. J Am Coll Cardiol. 2004 Nov 2;44(9):1780-5. doi: 10.1016/j.jacc.2004.07.043. PMID 15519007
- [Background] Adolph E, Holdt-Lehmann B, Chatterjee T, Paschka S, Prott A, Schneider H, Koerber T, Ince H, Steiner M, Schuff-Werner P, Nienaber CA. Renal Insufficiency Following Radiocontrast Exposure Trial (REINFORCE): a randomized comparison of sodium bicarbonate versus sodium chloride hydration for the prevention of contrast-induced nephropathy. Coron Artery Dis. 2008 Sep;19(6):413-9. doi: 10.1097/MCA.0b013e3283021ac6. PMID 18955835
- [Background] Marenzi G, Assanelli E, Marana I, Lauri G, Campodonico J, Grazi M, De Metrio M, Galli S, Fabbiocchi F, Montorsi P, Veglia F, Bartorelli AL. N-acetylcysteine and contrast-induced nephropathy in primary angioplasty. N Engl J Med. 2006 Jun 29;354(26):2773-82. doi: 10.1056/NEJMoa054209. PMID 16807414
- [Background] Tepel M, van der Giet M, Schwarzfeld C, Laufer U, Liermann D, Zidek W. Prevention of radiographic-contrast-agent-induced reductions in renal function by acetylcysteine. N Engl J Med. 2000 Jul 20;343(3):180-4. doi: 10.1056/NEJM200007203430304. PMID 10900277
- [Background] Chandel NS, McClintock DS, Feliciano CE, Wood TM, Melendez JA, Rodriguez AM, Schumacker PT. Reactive oxygen species generated at mitochondrial complex III stabilize hypoxia-inducible factor-1alpha during hypoxia: a mechanism of O2 sensing. J Biol Chem. 2000 Aug 18;275(33):25130-8. doi: 10.1074/jbc.M001914200. PMID 10833514
- [Background] DiMari J, Megyesi J, Udvarhelyi N, Price P, Davis R, Safirstein R. N-acetyl cysteine ameliorates ischemic renal failure. Am J Physiol. 1997 Mar;272(3 Pt 2):F292-8. doi: 10.1152/ajprenal.1997.272.3.F292. PMID 9087670
- [Background] Briguori C, Airoldi F, D'Andrea D, Bonizzoni E, Morici N, Focaccio A, Michev I, Montorfano M, Carlino M, Cosgrave J, Ricciardelli B, Colombo A. Renal Insufficiency Following Contrast Media Administration Trial (REMEDIAL): a randomized comparison of 3 preventive strategies. Circulation. 2007 Mar 13;115(10):1211-7. doi: 10.1161/CIRCULATIONAHA.106.687152. Epub 2007 Feb 19. PMID 17309916
- [Background] Solomon R, Deray G; Consensus Panel for CIN. How to prevent contrast-induced nephropathy and manage risk patients: practical recommendations. Kidney Int Suppl. 2006 Apr;(100):S51-3. doi: 10.1038/sj.ki.5000375. No abstract available. PMID 16612402
- [Background] McCullough PA, Wolyn R, Rocher LL, Levin RN, O'Neill WW. Acute renal failure after coronary intervention: incidence, risk factors, and relationship to mortality. Am J Med. 1997 Nov;103(5):368-75. doi: 10.1016/s0002-9343(97)00150-2. PMID 9375704
- [Background] Navaneethan SD, Singh S, Appasamy S, Wing RE, Sehgal AR. Sodium bicarbonate therapy for prevention of contrast-induced nephropathy: a systematic review and meta-analysis. Am J Kidney Dis. 2009 Apr;53(4):617-27. doi: 10.1053/j.ajkd.2008.08.033. Epub 2008 Nov 22. PMID 19027212
- [Background] Solomon R. The role of osmolality in the incidence of contrast-induced nephropathy: a systematic review of angiographic contrast media in high risk patients. Kidney Int. 2005 Nov;68(5):2256-63. doi: 10.1111/j.1523-1755.2005.00684.x. PMID 16221227
- [Background] Ozcan EE, Guneri S, Akdeniz B, Akyildiz IZ, Senaslan O, Baris N, Aslan O, Badak O. Sodium bicarbonate, N-acetylcysteine, and saline for prevention of radiocontrast-induced nephropathy. A comparison of 3 regimens for protecting contrast-induced nephropathy in patients undergoing coronary procedures. A single-center prospective controlled trial. Am Heart J. 2007 Sep;154(3):539-44. doi: 10.1016/j.ahj.2007.05.012. PMID 17719303
- [Derived] Leone AM, De Caterina AR, Sciahbasi A, Aurelio A, Basile E, Porto I, Trani C, Burzotta F, Niccoli G, Mongiardo R, Mazzari MA, Buffon A, Panocchia N, Romagnoli E, Lioy E, Rebuzzi AG, Crea F. Sodium bicarbonate plus N-acetylcysteine to prevent contrast-induced nephropathy in primary and rescue percutaneous coronary interventions: the BINARIO (BIcarbonato e N-Acetil-cisteina nell'infaRto mIocardico acutO) study. EuroIntervention. 2012 Nov 22;8(7):839-47. doi: 10.4244/EIJV8I7A127. PMID 23171803